CLINICAL TRIAL: NCT05256914
Title: Ozonized In-office and Domiciliary Gels vs Chlorhexidine Gel 1% for the Management of Peri-implant Mucositis Sites: a Randomized Clinical Trial.
Brief Title: Ozonized In-office and Domiciliary Gels vs Chlorhexidine Gel 1% for the Management of Peri-implant Mucositis Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-OZORAL6MONTHS
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Gels concealed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri-implant mucositis sites (Experimental): Peri-implant mucositis sites will be randomly assigned to ozone treatment.
  Interventions: Other: Ozoral Pro and Ozoral gel administration
- Contralateral peri-implant mucositis sites (Experimental): Contralateral peri-implant mucositis sites with respect to those treated with ozone will be assigned to chlorhexidine treatment.
  Interventions: Other: Curasept chlorhexidine gel 1%

INTERVENTIONS:
Other: Ozoral Pro and Ozoral gel administration — Peri-implant mucositis sites will receive in-office Ozoral Pro administration after non-surgical therapy. Patients will use Ozoral Gel for the domiciliary administration once a day for 14 days after the visits (no rinsing and eating for 30 minutes after gel application).
  Arms: Peri-implant mucositis sites
Other: Curasept chlorhexidine gel 1% — Peri-implant mucositis sites will receive in-office Curasept chlorhexidine gel 1% administration after non-surgical therapy. Patients will use chlorhexidine gel 1% for the domiciliary application once a day for 14 days after the visits (no rinsing and eating for 30 minutes after gel application).
  Arms: Contralateral peri-implant mucositis sites

SUMMARY:
This is a split-mouth randomized controlled clinical trial (RCT). After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with titanium curettes and air polishing with glycine powder.

After that, the following treatment will be randomly assigned:

* Ozoral Pro and Ozoral gel administration and home application for 2 peri-implant mucositis sites.
* Curasept chlorhexidine gel 1% administration and domiciliary application for 14 days for 2 peri-implant contralateral sites.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3). Professional hygiene will be performed again at T2 and T3.

At each recall session, the following periodontal clinical indices were collected using a probe on each peri-implant site: BOP, GBI, conditions of the marginal mucosa (swelling and erythema), suppuration, migration of the marginal mucosa, PD, PI ,BS.

DETAILED DESCRIPTION:
This is a split-mouth randomized controlled clinical trial (RCT). 30 patients is expected to be enrolled. After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with titanium curettes and air polishing with glycine powder.

After that, the following treatment will be randomly assigned:

* Ozoral Pro and Ozoral gel administration and home application for 2 peri-implant mucositis sites.
* Curasept chlorhexidine gel 1% administration and domiciliary application for 14 days for 2 peri-implant contralateral sites.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), and after 6 months (T3). At T2 and T3, professional hygiene will be performed again.

At each recall session, the following periodontal clinical indices were collected using a probe on each peri-implant site:

BOP (bleeding on probing) and GBI (gingival bleeding index) Conditions of the marginal mucosa (swelling and erythema) Suppuration Migration of the marginal mucosa PD (probing depth) PI (plaque index) BS (bleeding score)

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* presence of 2 peri-implant mucositis sites per side (left and right) with PD > 5 mm
* no systemic, metabolic and autoimmune disease
* compliant patients

Exclusion Criteria:

* neurologic, psychiatric and mental diseases
* patients taking bisphosphonates in the last 12 months
* patients taking antibiotics during the study
* pregnant and breastfeeding women
* patients undergoing anticancer treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Change in Bleeding on Probing (BOP%) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Dichotomous scoring (yes/no) of bleeding sites
Change in Gingival Bleeding Index (GBI%) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Quantitative assessment (percentage) of the bleeding sites (6 per tooth in total).
  Formula = n ° bleeding sites / n ° probed sites x100
Change in Suppuration (%) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Dichotomous scoring (yes/no) of suppurating sites
Change in marginal mucosa condition | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Scoring criteria:
  0: normal mucosa
  1. minimal inflammation with color change and minor edema
  2. moderate inflammation with redness, edema and glazing
  3. severe inflammation with redness, edema, ulceration and spontaneous bleeding without probing
Change in mucosal margin | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Dichotomous scoring (migrated/non migrated)
Change in Probing Depth (PD) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in Plaque Index (PI% - O' Leary Index) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
  Formula = n ° sites with plaque / total n ° of dental surfaces x100
Change in Bleeding Score (BS - Mombelli et al.) | Baseline (T0), after 1 (T1), 3 (T2) and 6 months (T3)
  Scoring criteria:
  0: no bleeding
  1. isolated visible spots
  2. blood forms a confluent red line on the mucosal margin
  3. profuse and copious bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data are available upon motivated request to the Authors.